CLINICAL TRIAL: NCT04599894
Title: Effect of Application of Low Dose of Pregabalin in TJA Before the Day of Surgery on Reducing Postoperative Side Effect of This Medicine
Brief Title: Reducing Postoperative Side Effect of Pregabalin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QiXin1
Record Dates: First submitted 2020-10-08; First posted 2020-10-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip
Keywords: pregabalin; total joint arthroplasty; side effect
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Sham Comparator): Oral administration of Pregabalin (75mg) 2h before operation; and oral administration of Pregabalin (75mg) at 18 pm from the first day after operation to discharge.
  Interventions: Drug: 75mg Pregabalin
- study group (Experimental): Oral administration of Pregabalin (37.5mg) at 8 am and 18 pm 1 d before operation; oral administration of Pregabalin (75mg) 2h before operation; and oral administration of Pregabalin (75mg) at 18 pm from the first day after operation to discharge.
  Interventions: Drug: 37.5mg Pregabalin + 75mg Pregabalin

INTERVENTIONS:
Drug: 37.5mg Pregabalin + 75mg Pregabalin — 37.5mg pregabalin preoperatively + 75mg pregabalin postoperatively
  Arms: study group
Drug: 75mg Pregabalin — 75mg pregabalin postoperatively
  Arms: control group

SUMMARY:
The purpose of this study was to determine 1) if pregabalin, when given 37.5 mg twice on the day before surgery, would be effective in reducing the early postoperative side effects including dizziness, nausea, vomiting and sedation of receiving pregabalin 75mg two hours pre-operatively and 75mg per day until the third postoperative day; and 2) whether this intervention affected the opioids consumption, and independent transfers at six hours post-op, time to readiness for independent transfers, time to readiness for discharge and pain or not.

DETAILED DESCRIPTION:
Study design This prospective randomized controlled clinical trial was conducted at our institution in accordance with the Declaration of Helsinki. The Institutional Review Board approved the study (IRB number IRB00008484). We registered the clinical trial on The ClinicalTrials.gov Protocol Registration (NCT04599894) before the enrolment of the first participant. Written informed consent was obtained from each patient.

Participant recruitment Patients were eligible for inclusion if they were between 18 and 80 years of age and scheduled for a primary TJA. Exclusion criteria included: medical history of neuropathic pain or other non-arthritic chronic pain; Non-steroidal anti-inflammatory drug intolerance or long-term use of opioids; psychiatric disorders; motion sickness.

Sample size estimation The sample size was based on a preliminary study (under the same synergy of medications, celecoxib (Pfizer) 400mg and pregabalin (Pfizer) 75mg two hours pre-operatively orally, on the day of surgery). The preliminary study demonstrated that only one patient fell dizziness postoperatively in ten consecutive TJA patients who received 37.5mg pregabalin twice on the day before surgery, while four patient fell dizziness postoperatively in ten consecutive TJA patients receiving none on the day before surgery. Therefore the sample size was calculated by comparing estimated proportion using the Chi-squared statistic, a sample size of 58 (29 per group) would reveal differences at the 5% level of significance, and with a power of 0.8.

Randomization A computer-generated randomization schedule was used to assign patients to one of two treatment groups. The schedule was created by the clinical research center of our hospital, which was not involved in the clinical care of patients or in the conduct of the present trial.

Treatment protocol All patients scheduled to undergo primary TJA between November 2020 and April 2021 were screened for recruitment. Participants were recruited at their preoperative assessment visit two days before surgery and were randomly assigned to one of two treatment groups. Group 1 (G1) received pregabalin 37.5 mg twice orally (PO) on the day before surgery (at 8 am and 6 pm, respectively), and celecoxib 400mg as well as pregabalin 75mg PO at two hours pre-operatively; Group 2 (G2) received none on the day before surgery and the same dose of celecoxib and pregabalin PO at two hours pre-operatively. Crystalloid for resuscitation was started on the morning of surgery. Perioperative antibiotics, cefazolin sodium, 2g, and tranexamic acid 1g were administered within one hour of skin incision via intravenous (IV) drip. Dolasetron 12.5mg IV and dexamethasone 5mg IV were administrated during the induction of anesthesia. Patients were sedated with midazolam and received a general anesthesia combined with fascia iliaca compartment block (FICB) for THA(0.2% ropivacaine 60mg for each joint) and adductor canal as well as infiltration between the popliteal Artery and Capsule of the Knee (iPACK) block for TKA (totally 0.2% ropivacaine 60mg for each joint). All procedures were performed by one group of surgeons (QX, GYH, ZXY, ZJT) through a posterolateral approach for THA and medial parapatellar approach for TKA. Periarticular injection (0.2% ropivacaine 80mg, compound betamethasone 7mg, ketorolac 30mg, epinephrine 0.3mg for each joint) was performed before implanting prosthesis. Cementless prosthesis (Depuy, Corail® Total Hip System) was used in all hips, and cemented prosthesis (Depuy, Attune® Total Knee System) was used in all knees. Neither drain was used in all wounds, nor was urinary catheter. IV patient-controlled analgesia (PCA) was not administered in these participants. Since two hours after extubation under general anesthesia, participants were allowed to drink water and progressively transit to their daily diaries. They were instructed to make independent postoperative transfers at six hours after extubation, which was taken as the final time point to determine the success of EARS pathway. Then these patients were transferred to a rehabilitation unit in the same hospital, cryotherapy and rehabilitation protocols were ordered until discharge. Rivaroxaban (10mg at 8 am per day, Bayer), celecoxib (200mg twice a day, at 8 am and 2 pm, respectively) as well as pregabalin (75mg per day at 6 pm) until the third postoperative day. Patients were instructed to maintain a VAS (visual analogous scale) pain score of between 1 and 3. If the VAS pain score was ≥4 at rest, oxycodone-acetaminophen (5mg/325mg, per dose, Mallinckrodt Inc.) would be used every six hours as needed for postoperative rescue analgesia. The discharge criteria included: patients' general well-being and acceptable pain control (VAS<4); dry wound; ability to safely mobilize with crutches and climb the stairs; patients' express acceptance of discharge; patients and family members learned the home-based exercise protocols for the first six weeks. Rivaroxaban was continued to use for five weeks. Cryotherapy, rehabilitation protocols and celecoxib 200mg twice a day were continued to use for six weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of knee osteoarthritis；
* avascular necrosis of femoral head；
* dysplasia of the hip joint.

Exclusion Criteria:

* medical history of neuropathic pain or other non-arthritic chronic pain;
* Non-steroidal anti-inflammatory drug intolerance or long-term use of opioids；
* psychiatric disorders;
* motion sickness.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
dizziness | at the night pre-operatively (at 8 pm)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | at two hours pre-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | at two hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | at four hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | at six hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | on the morning of postoperative day (POD) 1 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | on the morning of postoperative day (POD) 2 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
dizziness | on the morning of postoperative day (POD) 3 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)

SECONDARY OUTCOMES:
nausea | at the night pre-operatively (at 8 pm)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | at two hours pre-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | at two hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | at four hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | at six hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | on the morning of postoperative day (POD) 1 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | on the morning of postoperative day (POD) 2 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
nausea | on the morning of postoperative day (POD) 3 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | at the night pre-operatively (at 8 pm)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | at two hours pre-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | at two hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | at four hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | at six hours post-operatively
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | on the morning of postoperative day (POD) 1 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | on the morning of postoperative day (POD) 2 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
vomiting | on the morning of postoperative day (POD) 3 (at 8 am)
  assessed on a 4-point verbal rating scale (VRS) (none, mild, moderate and severe)
sedation | at the night pre-operatively (at 8 pm)
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | at two hours pre-operatively
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | at two hours post-operatively
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | at four hours post-operatively
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | at six hours post-operatively
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | on the morning of postoperative day (POD) 1 (at 8 am)
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | on the morning of postoperative day (POD) 2 (at 8 am)
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
sedation | on the morning of postoperative day (POD) 3 (at 8 am)
  ssessed by The Richmond Agitation-Sedation Scale (RASS)
opioids consumption | from surgery day to discharge day
  calculated as a product of the morphine equivalence and count, and intraoperative or any postoperative opioids consumption were recorded
independent transfers at six hours post-op | at six hours post-operatively
  calculated as a product of the morphine equivalence and count, and They were instructed to make safely independent postoperative transfers at six hours after extubation.
pain score | at six hours post-operatively
  Pain scores at rest and mobilization were assessed using VAS (0=no pain; 10=worst pain)
pain score | on the morning of postoperative day (POD) 1 (at 8 am)
  Pain scores at rest and mobilization were assessed using VAS (0=no pain; 10=worst pain)
pain score | on the morning of postoperative day (POD) 2 (at 8 am)
  Pain scores at rest and mobilization were assessed using VAS (0=no pain; 10=worst pain)
pain score | on the morning of postoperative day (POD) 3 (at 8 am)
  Pain scores at rest and mobilization were assessed using VAS (0=no pain; 10=worst pain)
time to readiness for discharge | from the day of independent transfers to the day of meeting discharge criteria
  Time to readiness for dischargey was calculated by day.
time to readiness for independent transfers | from the hour of extubation to the hour of independent transfers
  Time to readiness for dischargey was calculated by hour.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No